CLINICAL TRIAL: NCT02204280
Title: Urine UbA52 is a Biomarker of Early Diabetic Nephropathy
Brief Title: The Significance of Urine UbA52 In the Diagnosis of Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: Hebei Medical University Third Hospital (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: HebeiMUTH
Record Dates: First submitted 2014-07-23; First posted 2014-07-30 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Diabetic Nephropathy
Keywords: UbA52;diabetic nephropathy ;diabetic;ELISA
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — morning urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Type 2 Diabetic: Patiens with type 2 diabetic which conform to the WHO in 1999 diabetes diagnostic criteria.
- Diabetic With macro-or Microalbuminuria: Patients with diabetic with macro-or microalbuminuria.
- proteinuria,nondiabetic renal disease: Patients with proteinuria due to nondiabetic renal disease,such as IgA nephropathy,FSGS,Hypertensive renal damage and MN.
- healthy controls: Healthy person.

SUMMARY:
Definite diagnosis of diabetic nephropathy is currently based on renal biopsy findings. In most cases, however, the diagnosis can be reliably made in patients with macroalbuminuria in the presence of diabetic retinopathy.Microalbuminuria is often used as a prognostic marker in type 1 diabetes, because approximately 50% of type 1 diabetes patients with microalbuminuria will eventually develop diabetic nephropathy. Conversely, microalbu- minuria is of much less value as a marker in DM because it has a variety of causes, including hypertension. Thus, additional markers are needed to identify patient groups with a high risk of developing overt diabetic nephropathy. The aims of this study is checking urine UbA52 levels with ELISA to identify its significance in the diagnosis of diabetic nephropathy.

DETAILED DESCRIPTION:
It is now well recognized that the incidence of diabetes is increasing worldwide. It is the leading cause of end-stage renal disease (ESRD) in Western countries. Diabetic nephropathy has been reported to occur in 25%-40% of people with diabetes. The appearance of microalbuminuria usually is regarded as incipient nephropathy, but recently, work has suggested that some individuals with diabetes and decreased GFR may not have an increased urinary AER.Identification of markers for prediction of the clinical course of diabetic nephropathy remains a major challenge. Previous research showed that m/z14766 protein by mass spectrometry, was selectively excreted in the urine of diabetic nephropathy patients, the m/z 14766 mass peaks were identified as UbA52. We suppose that UbA52 can be regard as a simple and practical biomarker for diagnosis of diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. diabetes diagnostic criteria (WHO, 1999),age < 80 years old, gender not limited;
2. diabetic with macro-or microalbuminuria;
3. the subjects not took hemodialysis;
4. with proteinuria due to nondiabetic renal disease :Hypertensive renal damage,drug-induced acute interstitial nephritis, IgA, primary membranous nephropathy,FSGS or MCD, which were confirmed by renal biopsy.

Exclusion Criteria:

1. acute diabetic complications: ketoacidosis, hypertonic coma;
2. the diagnosis of malignant tumors, particularly affecting the liver and kidney function of tumor and the application of radiation and chemotherapy treatment of patients;
3. cardiac insufficiency, heart function class 3 or above;
4. data is not complete, have an impact on the results;
5. not hospitalized patients;
6. accept long-term oral or static point methods such as steroid hormone therapy, application of renal toxicity of drugs;
7. with the exception of primary kidney disease and other causes lead to eye disease;
8. the combination of respiratory system infection or other systemic diseases and patients with severe primary diseases, vigorous exercise within 24 hours;
9. pregnancy or breastfeeding women
10. there is a clear liver disease, its alanine or aspertate aminotransferase 2 times higher than normal limit;
11. reluctant to collaborators and psychiatric patients;
12. has been undergoing hemodialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with type 2 diabetic,diabetic with macro-or microalbuminuria and proteinuria due to nondiabetic renal disease from Hebei Medical University the Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The urine UbA52 levels in 30 patients with type 2 diabetic mellitus,30 patients with diabetic nephropathy，30 patients with proteinuria due to nondiabetic renal disease and 30 healthy persons | 12 months

REFERENCES:
- [Derived] Xu X, Dong Y, Liu M, Li Y, Zhang Y. Clinical significance of UbA52 level in the urine of patients with type 2 diabetes mellitus and diabetic kidney disease. Nefrologia (Engl Ed). 2021 Sep-Oct;41(5):548-555. doi: 10.1016/j.nefroe.2021.11.009. PMID 36165137